CLINICAL TRIAL: NCT06307392
Title: Bougie Versus Endotracheal Tube Alone on First-attempt Intubation Success in Prehospital Emergency Intubation in Patients Without Predictors of Difficult Intubation (BETA Trial)
Brief Title: Bougie Versus Endotracheal Tube Alone on First-attempt Intubation Success in Prehospital Emergency Intubation (BETA Trial)
Acronym: BETA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC22_0393
Record Dates: First submitted 2024-03-06; First posted 2024-03-12 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Failure Requiring Intubation
Keywords: Bougie; Intubation; Acute Respiratory failure; Airway; Critical Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endotracheal tube plus bougie (Experimental)
  Interventions: Procedure: First intubation attempt with endotracheal tube plus bougie
- Endotracheal tube alone (Active Comparator)
  Interventions: Procedure: First intubation attempt with endotracheal tube alone

INTERVENTIONS:
Procedure: First intubation attempt with endotracheal tube plus bougie — Use of a straight, malleable, semirigid bougie on first-attempt intubation. The required bougie is at least 60cm length, a coudé tip is recommended but not required. Operator may choose whether to bend the bougie prior to intubation.
  During laryngoscopy, the operator will insert the bougie into the trachea under direct or indirect visual control. If the bougie is successfully placed in the trachea, an assistant will load the endotracheal tube directly over the bougie while the operator will manually stabilize the bougie. Once the bougie has reached the mouth, the assistant will then stabilize the bougie, and the operator will advance the tube through the vocal cords to the adequate depth in the trachea, without removing the laryngoscope from the mouth. The operator will inflate the cuff and manually stabilize the tube. Then, the assistant will withdraw the bougie from the endotracheal tube.
  The use of a stylet is not permitted.
  Arms: Endotracheal tube plus bougie
Procedure: First intubation attempt with endotracheal tube alone — During laryngoscopy, the operator will insert the endotracheal tube alone into the trachea under direct or indirect visual control. The operator will advance the tube through the vocal cords to the adequate depth in the trachea, without removing the laryngoscope from the mouth. The operator will inflate the cuff and manually stabilize the tube.
  The use of a stylet is not permitted.
  Arms: Endotracheal tube alone

SUMMARY:
Emergency intubation is routinely performed in the prehospital setting. Airway management in the prehospital setting has substantial challenges, such as hostile environment or lack of technical support in case of first attempt intubation failure, and inherent risk of complications, such as hypoxemia, aspiration or oesophageal intubation. This risk is higher when several attempts are needed to succeed endotracheal intubation. Thus, a successful first attempt intubation is highly desirable to avoid adverse intubation-related events. Noteworthy, prehospital emergency intubation is associated with a lower rate of first attempt intubation success when compared to emergency intubation in the emergency department (ED). Research is needed to overcome the specific challenges of airway management in the prehospital setting, and to improve the safety and efficiency of prehospital emergency intubation. Literature reports that the use of assistive devices such as bougie may increase the rate of first-attempt intubation success in the ED. To date, no randomized trial has ever studied this device in the prehospital setting. Thus, the aim of the BETA trial is to compare first attempt intubation success facilitated by the bougie versus the endotracheal tube alone in the prehospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Managed by a physician staffed mobile intensive care unit (MICU).
* With an indication of emergency prehospital endotracheal intubation.

Exclusion Criteria:

* Pregnant women
* Patients with a "not to be resuscitated" indication.
* Patients with predictors of difficult intubation (that can be collected in the prehospital setting, including previous history of face, neck, throat surgery or pathology, limited mandibular protrusion, cervical spine trauma, facial trauma, ear-nose-throat malignancy, head or neck burns, history of previous difficult airways) for whom the use of a bougie is indicated on first intubation attempt.
* Patients under guardianship, trusteeship or safeguard of justice and patients with no health insurance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2027-03-26 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of first pass success during prehospital emergency intubation | Within 10 minutes following blade introduction
  Successful intubation on first attempt

SECONDARY OUTCOMES:
Occurrence of hypoxia | Within 1 hour following intubation
  SpO2 (pulsed oxygen saturation) <90%
Occurrence of bradycardia | Within 1 hour following intubation
  Heart rate <50 bpm
Occurrence of cardiac arrest | Within 1 hour following intubation
Occurrence of death | Within 1 hour following intubation
Occurrence of pulmonary aspirations | Within 1 hour following intubation
Occurrence of severe cardiovascular collapse | Within 1 hour following intubation
  Systolic blood pressure less than 65mmHg recorded at least once or less than 90 mmHg lasting 30 minutes despite 500-1,000 ml of fluid loading (crystalloids) or requiring introduction or increasing doses by more than 30% of vasoactive support
Time between blade introduction to the confirmation of a correct tube placement | Within 15 minutes following blade introduction
  In minutes. The correct position of the endotracheal tube is confirmed by detection of end-tidal carbon dioxide.
Change in SpO2 (pulsed oxygen saturation) from the time of induction to lowest SpO2 up to 2 minutes after confirmation of correct tube placement | Within 15 minutes following induction
  In percentage
Occurrence of change in SpO2 of more than 3% from the time of induction to 2 minutes after confirmation of correct tube placement | Within 15 minutes following induction
Cormack-Lehane grade of glottic view at first intubation attempt | Within 10 minutes following first blade introduction
Number of laryngoscopies attempts to achieve correct endotracheal tube placement | Within 30 minutes following first blade introduction
Number of patients for whom the placement of an endotracheal tube was not possible in the pre-hospital setting | Within 30 minutes following first blade introduction
Difficulty perceived by the operator on first intubation attempt | Within 10 minutes following blade introduction
  3-point Likert scale
Occurrence of injuries | Within 24 hours following intubation
  Occurrence (yes/no) of injuries related to the intubation:
  mucosal bleeding, laryngeal, tracheal, bronchial, mediastinal or oesophageal injuries
Occurrence of complications | Within 48 hours following intubation
  Occurrence (yes/no) of complications related to the intubation:
  aspiration pneumonia (new opacity on chest imaging within 48 hours after intubation, in comparison to the first chest imaging after hospital admission), pneumothorax (new air collection within the pleural cavity on chest imaging)
Change of SpO2/FiO2 ratio (pulsed oxygen saturation / fraction of inspired oxygen) between the time of confirmation of correct tube placement and the minimum ratio | Within one hour after confirmation of correct tube placement
  SpO2/FiO2 collected every 10 minutes to determine the minimum ratio

CONTACTS AND LOCATIONS:
Overall Officials: Quentin LE BASTARD, MD, Principal Investigator — Nantes University Hospital
Locations (10):
- France (10):
  - Nantes University Hospital, Nantes, Loire Atlantique
  - CHU de Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHD La Roche sur Yon, La Roche-sur-Yon
  - CH de Lorient, Lorient
  - CHU de Lyon, Lyon
  - CHU de Nancy, Nancy
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes

REFERENCES:
- [Derived] Le Bastard Q, Jenvrin J, Gaultier A, Montassier E. Bougie versus endotracheal tube alone on first-attempt intubation success in prehospital emergency intubation in patients without predictors of difficult intubation: protocol for the BETA randomized controlled trial. Trials. 2025 Sep 1;26(1):327. doi: 10.1186/s13063-025-09046-8. PMID 40890804